CLINICAL TRIAL: NCT05763992
Title: Targeting Triple Negative BREAst Cancer Metabolism With a Combination of Chemoimmunotherapy and a FASTing-like Approach in the Preoperative Setting: the BREAKFAST 2 Trial
Acronym: BREAKFAST-2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Collaborators: Istituto Oncologico Veneto IRCCS (Other); Ospedale Policlinico San Martino (Other); Federico II University (Other); Azienda Policlinico Umberto I (Other); European Institute of Oncology (Other); Ospedale "Carlo Poma" - Mantova (Other); Humanitas Clinical and Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INT214/22
Record Dates: First submitted 2023-01-18; First posted 2023-03-10 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2022-12

CONDITIONS: Breast Cancer; Triple Negative Breast Cancer; Dietary Exposure; Fasting
Keywords: Triple Negative Breast Cancer; Neoadjuvant chemoimmunotherapy; Fasting-Like Approach; Immunometabolism; Pathologic Complete Responses (pCRs); Randomized, phase II trial
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms; Fasting; Pathologic Complete Response

STUDY DESIGN:
Intervention Model Description: Multicenter, open-label, two-arm, comparative, randomized phase II study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Placebo Comparator): 12 consecutive cycles of weekly paclitaxel plus carboplatin (PCb) combined with 4 triweekly cycles of Pembrolizumab, followed by 4 consecutive cycles of triweekly anthracycline (doxorubicin or epirubicin)-cyclophosphamide (AC or EC) chemotherapy combined with 4 triweekly cycles of Pembrolizumab.
  Interventions: Dietary Supplement: Control diet (ARM A) or Fasting-Like Approach (FLA, ARM B)
- Arm B (Experimental): Standard treatment (12 consecutive cycles of weekly paclitaxel plus carboplatin (PCb) combined with 4 triweekly cycles of Pembrolizumab, followed by 4 consecutive cycles of triweekly anthracycline (doxorubicin or epirubicin)-cyclophosphamide (AC or EC) chemotherapy combined with 4 triweekly cycles of Pembrolizumab) in combination with up to a maximum of 8 consecutive triweekly cycles of 5-day Fasting-Like Approach
  Interventions: Dietary Supplement: Control diet (ARM A) or Fasting-Like Approach (FLA, ARM B)

INTERVENTIONS:
Dietary Supplement: Control diet (ARM A) or Fasting-Like Approach (FLA, ARM B) — Each FLA cycle will consist of 5 consecutive days of a specific FLA scheme, which will be repeated with a three-week interval. The FLA will consist of a plant-based, low-calorie (about 600 Kcal on day 1; about 300 Kcal on day 2 to 5), low-protein, low-carbohydrate diet. The first FLA cycle will start two days prior to the day of first chemo-immunotherapy cycle administration and will continue for two more days after chemotherapy. In the absence of significant contraindications or severe adverse events, subsequent FLA cycles will recur with three-week intervals and will maintain the same timing with respect to chemo-immunotherapy administration.

SUMMARY:
Italian, multicenter, open-label, two-arm, comparative, randomized phase II study investigating if the addition of the experimental metabolic intervention consisting in cycles of Fasting-Like Approach, as administered every three weeks up to a maximum of 8 consecutive cycles, is able to increase the anticancer activity of standard preoperative chemo-immunotherapy in patients with localized invasive Triple Negative Breast Cancer.

DETAILED DESCRIPTION:
TNBC is the most aggressive subtype of breast cancer. TNBC patients who achieve pCR during neoadjuvant chemo-immunotherapy have significantly lower rates of disease recurrence or death. Preclinical studies indicate that combining nutrient starvation, in the form of cycles of FLA, with anthracycline- or platinum-based chemotherapy remarkably increases the therapeutic index of chemotherapy against murine and human models of breast cancer, including models of TNBC. In particular, the chemotherapy-fasting/FLA combination increases the anticancer activity of chemotherapy, while reducing treatment-related adverse events (AEs). Moreover, the FLA has demonstrated potent and desirable immunomodulatory effects both in in vivo studies and in patients with cancer, and the activation of antitumor immunity is a crucial mediator of the anticancer effects of the FLA, either alone or in combination with chemotherapy. Therefore, there is a strong biological rationale to combine cyclic FLA with ICIs in cancer therapy.

Based on these data, we hypothesize that combining the FLA with standard-of-care, preoperative, anthracycline-taxane-carboplatin chemotherapy plus Pembrolizumab can increase the rate of pCR in a population of patients with stage II-III TNBC.

This is an Italian, multicenter, open-label, two-arm, comparative, randomized phase II study. This study is designed to investigate if the addition if the experimental metabolic intervention consisting in cycles of FLA, as administered every three weeks up to a maximum of 8 consecutive cycles, is able to increase the anticancer activity of standard preoperative chemo-immunotherapy consisting of antracycline-taxane-carboplatin-based chemotherapy plus pembrolizumab in patients with treatment naïve, localized (tumor stage T1c AND nodal stage N1-2, or tumor stage T2-4 AND nodal stage N0-2) invasive Triple Negative Breast Cancer (HER2 negative, ER <1%, PgR <1%). Bilateral and/or multifocal primary tumor is allowed, as well as inflammatory breast cancer, and the tumor with the most advanced T stage should be used to assess the eligibility. If multi-focal/multi-centric disease, TNBC needs to be confirmed for each focus. The primary study endpoint is pathologic complete response (pCR).

Patients will be randomly allocated to one of the following treatment arms:

* Arm A (control arm): 12 consecutive cycles of weekly paclitaxel plus carboplatin (PCb) combined with 4 triweekly cycles of Pembrolizumab, followed by 4 consecutive cycles of triweekly anthracycline (doxorubicin or epirubicin)-cyclophosphamide (AC or EC) chemotherapy combined with 4 triweekly cycles of Pembrolizumab. This combination treatment will be further referred to as "standard treatment".
* Arm B (experimental arm): standard treatment in combination with up to a maximum of 8 consecutive triweekly cycles of 5-day FLA.

Enrolled patients will be randomized in a 1:1 ratio and stratified according to a) disease stage: stage II (T1N1, T2N0, T2N1, T3N0) vs. stage III (T3N1; any T4; any N2); b) patient body mass index (BMI ≥25 kg/m2 vs <25 kg/m2).

After completion of the experimental preoperative protocol, patients will undergo surgery between 14 and 28 days after the last chemotherapy administration.

After surgery, patients will receive 9 additional triweekly pembrolizumab administration at the same dosage, and regardless of the pathologic tumor response (pCR yes vs. no). After surgery, patients may receive local radiotherapy, depending on the pathological stage and according to local and international guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Female sex
2. Age ≥ 18 and ≤ 75 years.
3. Evidence of a personally signed and dated informed consent document (ICD), signed and dated from the patient of legal representative with or without an impartial witness, indicating that the patient has been informed of all pertinent aspects of the study before enrollment
4. Willingness and ability to comply with the prescribed FLA regimen, the scheduled visits, treatment plans, laboratory tests and other procedures.
5. Histologically confirmed diagnosis of invasive TNBC candidate to neoadjuvant chemo-immunotherapy and subsequent curative surgery. On the basis of International Guidelines, TNBC is defined by absent or minimal (<1%) expression of oestrogen and progesterone receptors at IHC, and absence of HER2 protein over-expression and HER2 gene amplification, as defined as an IHC score of 0, 1+, or an IHC score of 2+ with in situ hybridization (ISH) analysis excluding HER2 gene amplification. The expression of hormone receptors (ER and PgR) and HER2 will be evaluated through immunohistochemistry (IHC), according to International Guidelines47,48
6. Availability of a formalin-fixed, paraffin-embedded (FFPE) block containing tumor tissue, or at least 7 unstained tumor slides.
7. Patients with tumor stage T1c AND nodal stage N1-2, or tumor stage T2-4 AND nodal stage N0-2 according to TNM.
8. Presence of an Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
9. Presence of adequate bone marrow and organ function as defined by the following laboratory values:

   1. ANC ≥ 1.5 x 103/l
   2. platelets ≥ 100 x 103/l
   3. hemoglobin ≥ 9.0 g/dl
   4. calcium (corrected for serum albumin) within normal limits or ≤ grade 1 according to NCI-CTCAE version 5.0 if not clinically significant
   5. potassium within the normal limits, or corrected with supplements
   6. creatinine < 1.5 ULN
   7. blood uric acid < 10 mg/dl
   8. ALT and AST ≤ 2 x ULN
   9. total bilirubin < 1.5 ULN except for patients with Gilbert syndrome who may only be included if the total bilirubin is < 3.0 x ULN or direct bilirubin < 1.5 x ULN
   10. Fasting glucose ≤ 250 mg/dl.
10. Female patients of childbearing potential must agree to sexual abstinence or to use two highly effective methods of contraception throughout the study and for at least six months after the end of the FLA. Abstinence is only acceptable if it is in line with the preferred and usual lifestyle of the patient. Examples of contraceptive methods with a failure rate of < 1% per year include tubal ligation, male sterilization, hormonal implants, established, proper use of combined oral or injected hormonal contraceptives, and certain intrauterine devices. Alternatively, two methods (e.g., two barrier methods such as a condom and a cervical cap) may be combined to achieve a failure rate of < 1% per year. Barrier methods must always be supplemented with the use of a spermicide. A patient is of childbearing potential if, in the opinion of the Investigator, she is biologically capable of having children and is sexually active.
11. Female patients are not of childbearing potential if they meet at least one of the following criteria:

    1. Have undergone a documented hysterectomy and/or bilateral oophorectomy
    2. Have medically confirmed ovarian failure
    3. Achieved post-menopausal status, defined as: ≥ 12 months of non-therapy-induced amenorrhea or surgically sterile (absence of ovaries); in women <45 years of age FSH level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy.

Exclusion Criteria:

1. Prior systemic treatment for breast cancer or other malignancies within 5 years of treatment enrollment, except for adequately treated basal cell or squamous skin cancer or in situ cervical cancer. Other malignancies diagnosed more than 5 years before the diagnosis of breast cancer must have been radically treated without evidence of relapse at the moment of patient enrollment in the trial.
2. Prior treatment with anthracyclines
3. Prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another co-inhibitory T-cell receptor (e.g., CTLA-4, OX-40, CD137)
4. Body mass index (BMI) < 19 kg/m2.
5. History of alcohol abuse.
6. Non-intentional weight loss ≥ 5% in the previous 3 months, unless the patient has a BMI > 22 kg/m2 and weight loss has been lower than 10% at the time of enrollment in the study; or non-intentional weight loss of ≥ 10% in the previous 3 months, unless the patient has a BMI > 25 kg/m2 and weight loss has been lower than 15% at the time of the enrollment in the study. In both cases, weight must have been stable for at least one month before study enrollment.
7. Active pregnancy or breast feeding.
8. Known active B or C hepatitis or human immunodeficiency virus (HIV) infection, or occasional finding of active hepatitis B/C infection during screening tests before chemotherapy initiation, as defined as positive polymerase chain reaction (PCR) testing for HBV-DNA and HCV-RNA and qualitative PCR for HIV-RNA, or requiring active treatment at study enrollment.
9. Serious infections in the previous 4 weeks before the FLA initiation, including, but not limited to, potential hospitalizations for complications of infections, bacteriemia or serious pneumonitis.
10. Active autoimmune diseases requiring systemic treatments (e.g., systemic steroids or immune suppressants). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment.
11. Active chronic therapy with systemic steroids at a dose ≥ 10 mg per day of prednisone or equivalent at study enrollment.
12. Diagnosis of type 1 or 2 diabetes mellitus requiring pharmacologic therapy (including, but not limited to, insulin or insulin secretagogues), with the exception of metformin. A diagnosis of type 2 diabetes mellitus not requiring pharmacological treatments, or only requiring treatment with metformin, based on the judgment of a diabetologist, is compatible with patient enrollment in the trial.
13. Anamnesis of clinically significant heart disease including:

    1. angina pectoris, coronary bypass, symptomatic pericarditis, myocardial infarction in the previous 12 months from the beginning of experimental therapy;
    2. congestive heart failure (NYHA III-IV).
14. Anamnesis of clinically meaningful cardiac arrhythmias, such as ventricular tachycardia, chronic atrial fibrillation, complete bundle branch block, high grade atrio-ventricular block like bi-fascicular block, type II Mobitz and third grade atrio-ventricular block, nodal arrhythmias, supra-ventricular arrhythmia.
15. Left ventricular ejection fraction lower than 50% at the cardiac scan with radionuclides or at echocardiography.
16. Previous episodes of symptomatic hypotension leading to loss of consciousness.
17. History of eating disorders (anorexia, bulimia).
18. Baseline plasma fasting glucose ≤ 60 mg/dL.
19. Medical or psychiatric comorbidities rendering the patient not candidate to the clinical trial, according to the investigator's judgement.
20. Other cardiac, liver, lung or renal comorbidities, not specified in the previous inclusion or exclusion criteria, but potentially exposing the patient to a high risk of lactic acidosis.
21. Known history of active TB (Bacillus Tuberculosis).

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Estimated)
Dates: Start 2023-05-15 (Estimated); Primary Completion 2025-05-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Rate of Pathologic complete response (pCR) | Surgical specimen (at the time of surgery)
  Absence of residual tumor cells in both breast tissue and axillary lymph nodes (ypT0/ypTis ypN0)

SECONDARY OUTCOMES:
Disease free survival (DFS) | Time from surgery to tumor recurrence or patient death, assessed up to 36 months
  Time from surgery to tumor recurrence, either local or distant, or patient death from any cause, assessed up to 36 months
Event-free survival (EFS) | From the date of randomization to the first documentation of progressive disease or patient death, assessed up to 36 months
  Time from the date of randomization to the first documentation of progressive disease, or patient death from any cause, assessed up to 36 months
Distant metastasis free survival (DMFS) | From surgery to the occurrence of distant metastases or patient death, assessed up to 36 months
  Time from surgery to the occurrence of distant metastases or patient death from any cause, assessed up to 36 months
Overall Survival (OS) | Time from randomization to the date of death, assessed up to 60 months
  Time from randomization to the date of death (patients alive at the time of data cut-off and analysis will be censored at their last contact date), assessed up to 60 months
Compliance (Dose-intensity) | From the start to the end of the neoadjuvant treatment (about 6 months)
  Dose of effective drug administrated per unit of time (e.g., mg/m2/week)
Compliance (Drug dose/time modifications) | From the start to the end of the neoadjuvant treatment (about 6 months)
  Percentage of patients with drug dose and/or time modifications
Compliance (Dietary regimen modifications) | From the start to the end of the neoadjuvant treatment (about 6 months)
  Percentage of patients with experimental dietary regimen modifications
Compliance (Withdrawals) | From the start to the end of the neoadjuvant treatment (about 6 months)
  Percentage of premature withdrawals
Safety (AE) | From the start to the end of the neoadjuvant treatment (about 6 months)
  Incidence, nature, severity and seriousness of AEs, according of NCI-CTCAE, version 5.0
Safety (Maximum toxicity grade) | From the start to the end of the neoadjuvant treatment (about 6 months)
  Maximum toxicity grade experienced by each patient for each specific toxicity
Safety (G3-G4 AEs) | From the start to the end of the neoadjuvant treatment (about 6 months)
  Percentage of patients experiencing grade 3-4 toxicity for each specific toxicity
Safety (SAE) | From the start to the end of the neoadjuvant treatment (about 6 months)
  Patients with at least a SAE

OTHER OUTCOMES:
Translational (DNA repair, metabolic, autophagy and immunologic parameters effect on pCR) | Surgical specimen (at the time of surgery)
  Role of key DNA repair, metabolic, autophagy and immunologic pathways in the efficacy of the experimental treatments, defined as the rate of pCR

CONTACTS AND LOCATIONS:
Overall Officials: Maria Vittoria Dieci, MD, Principal Investigator — Istituto Oncologico Veneto, Via Gattamelata 64, 35128 Padova, Italy; Matteo Lambertini, MD, Principal Investigator — IRCCS Ospedale Policlinico San Martino, Largo Rosanna Benzi 10, 16132 Genova; Sabino De Placido, MD, Principal Investigator — University of Naples Federico II, Via Sergio Pansini 5, 80131 Naples; Monica Iorfida, MD, Principal Investigator — Istituto Europeo di Oncologia; Alberto Zambelli, MD, Principal Investigator — Humanitas Research Hospital, Via Alessandro Manzoni 56, 20089 Rozzano; Andrea Botticelli, MD, Principal Investigator — "Sapienza" University of Rome, 00185, Rome; Carla Strina, MD, Principal Investigator — A.O. "Istituti Ospitalieri", Viale Concordia 1, 26100 Cremona
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kassam F, Enright K, Dent R, Dranitsaris G, Myers J, Flynn C, Fralick M, Kumar R, Clemons M. Survival outcomes for patients with metastatic triple-negative breast cancer: implications for clinical practice and trial design. Clin Breast Cancer. 2009 Feb;9(1):29-33. doi: 10.3816/CBC.2009.n.005. PMID 19299237
- [Result] Cortazar P, Zhang L, Untch M, Mehta K, Costantino JP, Wolmark N, Bonnefoi H, Cameron D, Gianni L, Valagussa P, Swain SM, Prowell T, Loibl S, Wickerham DL, Bogaerts J, Baselga J, Perou C, Blumenthal G, Blohmer J, Mamounas EP, Bergh J, Semiglazov V, Justice R, Eidtmann H, Paik S, Piccart M, Sridhara R, Fasching PA, Slaets L, Tang S, Gerber B, Geyer CE Jr, Pazdur R, Ditsch N, Rastogi P, Eiermann W, von Minckwitz G. Pathological complete response and long-term clinical benefit in breast cancer: the CTNeoBC pooled analysis. Lancet. 2014 Jul 12;384(9938):164-72. doi: 10.1016/S0140-6736(13)62422-8. Epub 2014 Feb 14. PMID 24529560
- [Result] Sikov WM, Berry DA, Perou CM, Singh B, Cirrincione CT, Tolaney SM, Kuzma CS, Pluard TJ, Somlo G, Port ER, Golshan M, Bellon JR, Collyar D, Hahn OM, Carey LA, Hudis CA, Winer EP. Impact of the addition of carboplatin and/or bevacizumab to neoadjuvant once-per-week paclitaxel followed by dose-dense doxorubicin and cyclophosphamide on pathologic complete response rates in stage II to III triple-negative breast cancer: CALGB 40603 (Alliance). J Clin Oncol. 2015 Jan 1;33(1):13-21. doi: 10.1200/JCO.2014.57.0572. Epub 2014 Aug 4. PMID 25092775
- [Result] Poggio F, Tagliamento M, Ceppi M, Bruzzone M, Conte B, Fregatti P, Punie K, de Azambuja E, Del Mastro L, Lambertini M. Adding a platinum agent to neoadjuvant chemotherapy for triple-negative breast cancer: the end of the debate. Ann Oncol. 2022 Mar;33(3):347-349. doi: 10.1016/j.annonc.2021.11.016. Epub 2021 Nov 30. No abstract available. PMID 34861375
- [Result] Cortes J, Cescon DW, Rugo HS, Nowecki Z, Im SA, Yusof MM, Gallardo C, Lipatov O, Barrios CH, Holgado E, Iwata H, Masuda N, Otero MT, Gokmen E, Loi S, Guo Z, Zhao J, Aktan G, Karantza V, Schmid P; KEYNOTE-355 Investigators. Pembrolizumab plus chemotherapy versus placebo plus chemotherapy for previously untreated locally recurrent inoperable or metastatic triple-negative breast cancer (KEYNOTE-355): a randomised, placebo-controlled, double-blind, phase 3 clinical trial. Lancet. 2020 Dec 5;396(10265):1817-1828. doi: 10.1016/S0140-6736(20)32531-9. PMID 33278935
- [Result] Mittendorf EA, Zhang H, Barrios CH, Saji S, Jung KH, Hegg R, Koehler A, Sohn J, Iwata H, Telli ML, Ferrario C, Punie K, Penault-Llorca F, Patel S, Duc AN, Liste-Hermoso M, Maiya V, Molinero L, Chui SY, Harbeck N. Neoadjuvant atezolizumab in combination with sequential nab-paclitaxel and anthracycline-based chemotherapy versus placebo and chemotherapy in patients with early-stage triple-negative breast cancer (IMpassion031): a randomised, double-blind, phase 3 trial. Lancet. 2020 Oct 10;396(10257):1090-1100. doi: 10.1016/S0140-6736(20)31953-X. Epub 2020 Sep 20. PMID 32966830
- [Result] Schmid P, Cortes J, Pusztai L, McArthur H, Kummel S, Bergh J, Denkert C, Park YH, Hui R, Harbeck N, Takahashi M, Foukakis T, Fasching PA, Cardoso F, Untch M, Jia L, Karantza V, Zhao J, Aktan G, Dent R, O'Shaughnessy J; KEYNOTE-522 Investigators. Pembrolizumab for Early Triple-Negative Breast Cancer. N Engl J Med. 2020 Feb 27;382(9):810-821. doi: 10.1056/NEJMoa1910549. PMID 32101663
- [Result] Gong Y, Ji P, Yang YS, Xie S, Yu TJ, Xiao Y, Jin ML, Ma D, Guo LW, Pei YC, Chai WJ, Li DQ, Bai F, Bertucci F, Hu X, Jiang YZ, Shao ZM. Metabolic-Pathway-Based Subtyping of Triple-Negative Breast Cancer Reveals Potential Therapeutic Targets. Cell Metab. 2021 Jan 5;33(1):51-64.e9. doi: 10.1016/j.cmet.2020.10.012. Epub 2020 Nov 11. PMID 33181091
- [Result] Vernieri C, Casola S, Foiani M, Pietrantonio F, de Braud F, Longo V. Targeting Cancer Metabolism: Dietary and Pharmacologic Interventions. Cancer Discov. 2016 Dec;6(12):1315-1333. doi: 10.1158/2159-8290.CD-16-0615. Epub 2016 Nov 21. PMID 27872127
- [Result] Salvadori G, Zanardi F, Iannelli F, Lobefaro R, Vernieri C, Longo VD. Fasting-mimicking diet blocks triple-negative breast cancer and cancer stem cell escape. Cell Metab. 2021 Nov 2;33(11):2247-2259.e6. doi: 10.1016/j.cmet.2021.10.008. PMID 34731655
- [Result] Caffa I, Spagnolo V, Vernieri C, Valdemarin F, Becherini P, Wei M, Brandhorst S, Zucal C, Driehuis E, Ferrando L, Piacente F, Tagliafico A, Cilli M, Mastracci L, Vellone VG, Piazza S, Cremonini AL, Gradaschi R, Mantero C, Passalacqua M, Ballestrero A, Zoppoli G, Cea M, Arrighi A, Odetti P, Monacelli F, Salvadori G, Cortellino S, Clevers H, De Braud F, Sukkar SG, Provenzani A, Longo VD, Nencioni A. Fasting-mimicking diet and hormone therapy induce breast cancer regression. Nature. 2020 Jul;583(7817):620-624. doi: 10.1038/s41586-020-2502-7. Epub 2020 Jul 15. PMID 32669709
- [Result] Di Tano M, Raucci F, Vernieri C, Caffa I, Buono R, Fanti M, Brandhorst S, Curigliano G, Nencioni A, de Braud F, Longo VD. Synergistic effect of fasting-mimicking diet and vitamin C against KRAS mutated cancers. Nat Commun. 2020 May 11;11(1):2332. doi: 10.1038/s41467-020-16243-3. PMID 32393788
- [Result] Vernieri C, Ligorio F, Zattarin E, Rivoltini L, de Braud F. Fasting-mimicking diet plus chemotherapy in breast cancer treatment. Nat Commun. 2020 Aug 26;11(1):4274. doi: 10.1038/s41467-020-18194-1. PMID 32848145
- [Result] Vernieri C, Fuca G, Ligorio F, Huber V, Vingiani A, Iannelli F, Raimondi A, Rinchai D, Frige G, Belfiore A, Lalli L, Chiodoni C, Cancila V, Zanardi F, Ajazi A, Cortellino S, Vallacchi V, Squarcina P, Cova A, Pesce S, Frati P, Mall R, Corsetto PA, Rizzo AM, Ferraris C, Folli S, Garassino MC, Capri G, Bianchi G, Colombo MP, Minucci S, Foiani M, Longo VD, Apolone G, Torri V, Pruneri G, Bedognetti D, Rivoltini L, de Braud F. Fasting-Mimicking Diet Is Safe and Reshapes Metabolism and Antitumor Immunity in Patients with Cancer. Cancer Discov. 2022 Jan;12(1):90-107. doi: 10.1158/2159-8290.CD-21-0030. Epub 2021 Nov 17. PMID 34789537
- [Result] Ligorio F, Fuca G, Provenzano L, Lobefaro R, Zanenga L, Vingiani A, Belfiore A, Lorenzoni A, Alessi A, Pruneri G, de Braud F, Vernieri C. Exceptional tumour responses to fasting-mimicking diet combined with standard anticancer therapies: A sub-analysis of the NCT03340935 trial. Eur J Cancer. 2022 Sep;172:300-310. doi: 10.1016/j.ejca.2022.05.046. Epub 2022 Jul 8. PMID 35810555

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-01): https://cdn.clinicaltrials.gov/large-docs/92/NCT05763992/Prot_SAP_000.pdf